CLINICAL TRIAL: NCT02698605
Title: Design and Usability Evaluation of a Novel Robotic Bilateral Arm Rehabilitation Device for Patients With Stroke
Brief Title: Evaluation of the Arm Rehabilitation Device for Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Alice May-Kuen Wong, Attending physician, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 101-5038A3
Record Dates: First submitted 2016-02-13; First posted 2016-03-03 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Usability test study of the MirrorPath (Experimental): This study was a one-arm study and all subjects used the device and received usability test.
  Interventions: Device: Usability test study of the MirrorPath

INTERVENTIONS:
Device: Usability test study of the MirrorPath — The study was conducted by research assistants. Each subject received one assessment that last lasted 30 minutes. The subjects were not paid for participation. In that, no randomization or masking were performed. Prior to the experiment part of the study, the subjects provided basic biographical information. We then explained the experimental process and demonstrated the operation of the device.
  A novel rehabilitation device, the MirrorPath, designed for the upper limb rehabilitation of patients with hemiplegic stroke. The MirrorPath that was 1180x440x300mm in size and had a shell was constructed of acrylonitrile butadiene styrene (ABS). The control module featured an on/off switch, a knob for adjusting the speed, and an emergency cutoff switch.

SUMMARY:
The usability assessment focuses on the actual use of the proposed rehabilitation system to clarify issues users would face in actual system operation, thus providing a reference for subsequent system improvement.

DETAILED DESCRIPTION:
This study protocol was approved by the institutional review board of Chang Gung Medical Foundation. The usability assessment focuses on the actual use of the proposed rehabilitation system to clarify issues users would face in actual system operation, thus providing a reference for subsequent system improvement. Pre-testing and formal testing were conducted at Chang Gung Memorial Hospital at Taoyuan. The pre-test was conducted on five healthy participants, while the formal testing was conducted on 12 participants (4 stroke patients, 4 caregivers, and 4 therapists). The healthy participants were aged 20-70 years old and had no physical disabilities; the stroke patients had normal cognitive and language skills, stable stroke status, no fractures in the upper limbs in the previous three months, and minimal or no upper limb spasticity with Modified Ashworth Scale of 0 or 1; the occupational therapists should had work experience in the hospital for more than one year.

Prior to the experiment, the subject provided basic biographical information. The investigators then explained the experimental process and demonstrated the operation of the device. For usability assessment, the subject operated the device under the instruction by the researchers, during which problems observed and questions asked were recorded. Following device operation, the subjects filled the system usability scale (SUS) questionnaire that obtained subjective evaluations and recommendations for the device. Experimental instrument consisted of the rehabilitation device, video cameras, still image cameras, digital voice recorders, questionnaires and observational recording forms.

The results of the SUS questionnaire were analyzed using SPSS (IBM Corp., Armonk, NY, USA). The split-half method was used for reliability analysis and one-sample t test for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Had previous experience using rehabilitation equipment.

Exclusion Criteria:

* Cognitive deficits or psychiatric illness.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The system usability scale (SUS) | Up to 2 year
  Up to twenty subjects with their age ranging from 20 years to 70 years are planned to recruit for the one-time SUS. Categorizing the SUS questionnaire items in relation to usability (Q1, Q2, Q3, Q5, Q6, Q7, Q8, Q9) and learning (Q4, Q10) domains.

CONTACTS AND LOCATIONS:
Overall Officials: Alice M Wong, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pei YC, Chen JL, Wong AMK, Tseng KC. An Evaluation of the Design and Usability of a Novel Robotic Bilateral Arm Rehabilitation Device for Patients with Stroke. Front Neurorobot. 2017 Jul 28;11:36. doi: 10.3389/fnbot.2017.00036. eCollection 2017. PMID 28804454